CLINICAL TRIAL: NCT03217812
Title: A Phase 3, Multicenter, Randomized, Controlled, Open-label Study of VELCADE (Bortezomib) Melphalan-Prednisone (VMP) Compared to Daratumumab in Combination With VMP (D-VMP), in Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High-Dose Therapy (Asia Pacific Region)
Brief Title: A Study of VELCADE (Bortezomib) Melphalan-Prednisone (VMP) Compared to Daratumumab in Combination With VMP (D-VMP), in Participants With Previously Untreated Multiple Myeloma Who Are Ineligible for High-Dose Therapy (Asia Pacific Region)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108340; 54767414MMY3011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-07-13; First posted 2017-07-14 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A: VMP Alone (Active Comparator): Participants will receive Velcade (bortezomib) 1.3 milligram per square meter (mg/m^2) as subcutaneous (SC) injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2 (if serum creatine is greater than [>]2 milligram per deciliter [mg/dL] at baseline, participants must be administrated 4.5 mg/m^2 of melphalan, instead of 9 mg/m^2) orally, once daily (on Days 1 to 4) and prednisone 60 mg/m^2, orally, once daily on Days 1 to 4 of each cycle up to Cycle 9.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone
- Treatment B: D-VMP (Experimental): Participants will receive Velcade 1.3 mg/m^2 as SC injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9, melphalan 9 mg/m^2 (if serum creatine is >2 mg/dL at baseline, participants must be administrated 4.5 mg/m^2 of melphalan, instead of 9 mg/m^2), orally, once daily (on Days 1-4) and prednisone 60 mg/m^2, orally, once daily, on Days 1 to 4 of each cycle up to Cycle 9. In addition participants will also receive daratumumab 16 milligram per kilogram (mg/kg) as intravenous (IV) infusion or daratumumab Subcutaneously (SC) at the discretion of the investigator, once weekly, for 6 weeks in Cycle 1 and then every 3 weeks, in Cycles 2 to 9 and thereafter, once every 4 weeks until documented progression, unacceptable toxicity, or the end of study. Participants will receive pre-infusion medications before each daratumumab infusion.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone; Drug: Daratumumab

INTERVENTIONS:
Drug: Velcade — Participants will receive velcade 1.3 mg/m^2, SC injection, twice weekly at Weeks 1, 2, 4 and 5 in Cycle 1 followed by once weekly at Weeks 1, 2, 4 and 5 in Cycles 2 to 9 of Treatment Arm A and B.
  Other Names: Bortezomib
Drug: Melphalan — Participants will receive melphalan 9 mg/m^2 (if serum creatine is >2 mg/dL at baseline, participants must be administrated 4.5 mg/m^2 of melphalan, instead of 9 mg/m^2), orally, once daily on Days 1 to 4 of each cycle up to Cycle 9 Treatment Arm A and B.
Drug: Prednisone — Participants will receive prednisone 60 mg/m^2, orally, once daily, on Days 1 to 4 of each cycle up to Cycle 9 Treatment Arm A and B.
Drug: Daratumumab — Participants will receive daratumumab 16 mg/kg as IV infusion or daratumumab SC, once weekly, for 6 weeks in Cycle 1 and then once every 3 weeks, in Cycle 2 to 9 and thereafter, once every 4 weeks until documented progression, unacceptable toxicity, or the end of study in Treatment Arm B.
  Other Names: JNJ-54767414
  Arms: Treatment B: D-VMP

SUMMARY:
The purpose of this study is to determine if the addition of daratumumab to VELCADE-melphalan-prednisone (VMP) will improve very good partial response (VGPR) or better compared with VMP alone.

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma satisfying the calcium elevation, renal insufficiency, anemia, and bone abnormalities (CRAB) diagnostic criteria, monoclonal plasma cells in the bone marrow greater than or equal to (>=) 10 percent (%) or presence of a biopsy proven plasmacytomas, and measurable secretory disease, as assessed by the central laboratory, and defined in protocol
* Newly diagnosed and not considered candidate for high-dose chemotherapy with stem cell transplantation (SCT) due to: being age >= 65 years, or in participants less than (<) 65 years: presence of important comorbid conditions likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Meet the clinical laboratory criteria as specified in the protocol
* A woman of childbearing potential must have a negative serum or urine pregnancy tests at screening within 14 days prior to randomization

Exclusion Criteria:

* Primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma
* Waldenstrom's disease, or other conditions in which Immunoglobulin M (IgM) M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Prior or current systemic therapy or SCT for multiple myeloma, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 milligram per day (mg/day) for 4 days) of corticosteroids before treatment
* Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the national cancer institute common terminology criteria for adverse events (NCI-CTCAE), Version 4.03
* History of malignancy (other than multiple myeloma) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years)
* Radiation therapy within 14 days of randomization
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (that is, participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [Anti-HBc] and/or antibodies to hepatitis B surface antigen [Anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. EXCEPTION: Participants with serologic findings suggestive of HBV vaccination (Anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Rate at 6 Month After Last Participant First Dose | At 6 months after last participant first dose (approximately up to 2.5 years)
  The VGPR or better rate, defined as the proportion of participants achieving VGPR and complete response (CR) (including stringent complete response [sCR]) according to the international myeloma working group (IMWG) criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than equal to (>=) 90 percent (%) reduction in serum M-protein plus urine M-protein <100 milligram (mg)/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and less than (<) 5% plasma cells (PCs) in bone marrow. sCR: CR plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.
Very Good Partial Response (VGPR) or Better Rate at 3 Years After Last Participant First Dose | At 3 years after last participant first dose (approximately up to 5 years)
  The VGPR or better rate, defined as the proportion of participants achieving VGPR and CR (including sCR) according to the IMWG criteria during or after the study treatment. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90 % reduction in serum M-protein plus urine M-protein <100 mg/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PCs) in bone marrow. sCR: CR plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  The PFS is defined as time from date of randomization to either Progressive disease (PD), death, whichever occurs first according to IMWG criteria. IMWG criteria for PD: Increase of 25% from lowest response value in any one of following: Serum M-component (absolute increase must be >=0.5 gram per deciliter (g/dL), Urine M-component (absolute increase must be >=200 mg/24 hours), Participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be >10 milligrams per deciliter (mg/dL), participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC% (absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia (serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time to Next Treatment | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Time to next treatment is defined as the time from randomization to the start of the next-line treatment.
Overall Response Rate (ORR) | At 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  The ORR is defined as the proportion of participants who achieve partial response (PR) or better according to IMWG criteria, during or after study treatment. IMWG criteria: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to <200 mg/24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Complete Response Rate | At 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Complete response based on IMWG criteria is defined as: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% PCs in bone marrow.
Stringent Complete Response (sCR) Rate | At 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Time to response, defined as the time between randomization and the first efficacy evaluation that the participant has met all criteria for PR or better. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by>=90% or to <200 mg/24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Time to Response | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Time to response, defined as the time between randomization and the first efficacy evaluation that the participant has met all criteria for PR or better. IMWG criteria for PR: >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by>=90% or to <200 mg/24 hours, If the serum and urine M-protein are not measurable, a decrease of >=50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria, If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow PCs is required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%. In addition to the above criteria, if present at baseline, a >=50% reduction in the size of soft tissue plasmacytomas is also required.
Overall Survival (OS) | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  The OS is defined as the time from the date of randomization to the date of the participant's death.
Duration of Response | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Duration of response is time from the date of initial documentation of response (PR or better) to the date of first documented evidence of PD, as defined by IMWG criteria. IMWG criteria for PD: Increase of 25% from lowest response value in any one of the following: Serum M-component (absolute increase must be >=0.5 g/dL, Urine M-component (absolute increase must be >=200 mg/24 hours), Participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be >10 milligram per deciliter (mg/dL), participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC%(absolute percentage must be >=10%), definite development of new bone lesions or soft tissue plasmacytomas or increase in size of bone lesions or tissue plasmacytomas and development of hypercalcemia ( serum calcium >11.5 mg/dL) that can be attributed solely to PC proliferative disorder.
Time to VGPR or Better Response | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Time to VGPR or better response defined as the time between randomization and the first efficacy evaluation that the participant has met all criteria for VGPR or better in responders. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than equal to (>=) 90 percent (%) reduction in serum M-protein plus urine M-protein <100 milligram (mg)/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PCs) in bone marrow. sCR: CR plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.
Duration of VGPR or Better Response | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Duration of VGPR or better response is calculated from the date of initial documentation of the first (VGPR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than equal to (>=) 90 percent (%) reduction in serum M-protein plus urine M-protein <100 milligram (mg)/24 hours, CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas and <5% plasma cells (PCs) in bone marrow. sCR: CR plus normal free light chain (FLC) ratio, and absence of clonal PCs by immunohistochemistry (IHC), immunofluorescence or 2- to 4 color flow cytometry.
EuroQoL 5-Dimension 5-Level Health Status (EQ-5D-5L) Questionnaire | At 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Health Status (QLQ-C30) Questionnaire | At 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  The EORTC QLQ-C30 includes 30 items resulting in 5 functional scales (physical, role, cognitive, emotional, and social), 1 global health status scale, 3 symptom scales (fatigue, pain, nausea/vomiting) and 6 single items (dyspnea, appetite loss, insomnia, constipation/diarrhea and financial difficulties). The recall period is 1 week (the past week). Scores are transformed to a 0 to 100 scale. Higher score=better level of functioning or greater degree of symptoms.
Number of Participants With Antibodies to Daratumumab | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Number of participants with antibodies to daratumumab will be analysed.
Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Clinical Efficacy of D-VMP in High Risk Molecular Subgroups | Up to 6 months after last participant first dose (approximately up to 2.5 years) and 3 years after last participant first dose (approximately up to 5 years)
  Clinical efficacy will be analyzed in high risk molecular subgroups between DVMP and VMP.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (43):
- China (29):
  - Beijing Chaoyang Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital, Central South University, Changsha
  - West China Hospital Si Chuan University, Chengdu
  - Second Affiliated Hospital of Army Medical University, Chongqing
  - Fujian Meidical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Nanfang Hospital, Guangzhou
  - First Affiliated Hospital Medical School of Zhejiang University, Hangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Changzheng Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - First Affiliated Hospital SooChow University, Suzhou
  - Tianjin cancer hospital, Tianjin
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - Tangdu Hospital, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Queen Mary Hospital University of Hong Kong, Hong Kong, Hong Kong
- Malaysia (3):
  - Hospital Ampang, Ampang
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
- South Korea (7):
  - Inje University Busan Paik Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Fu W, Bang SM, Huang H, Kim K, Li W, An G, Lee JJ, Cai Z, Jin J, Wang Y, Chim CS, Carson R, Liu R, Zhao M, Chen X, Cui C, Hou J, Wang J. Health-related quality of life with daratumumab, bortezomib, melphalan, and prednisone versus bortezomib, melphalan, and prednisone alone in transplant-ineligible patients with newly diagnosed multiple myeloma: analysis of the phase 3 OCTANS study. Ann Hematol. 2025 May;104(5):2765-2776. doi: 10.1007/s00277-025-06303-3. Epub 2025 May 23. PMID 40407887
- [Derived] Fu W, Bang SM, Huang H, Kim K, Li W, An G, Lee JJ, Cai Z, Jin J, Wang Y, Chim CS, Carson R, Liu R, Zhao M, Chen X, Cui C, Hou J, Wang J. Daratumumab, bortezomib, melphalan, and prednisone versus bortezomib, melphalan, and prednisone alone in transplant-ineligible Asian patients with newly diagnosed multiple myeloma: final analysis of the phase 3 OCTANS Study. Ann Hematol. 2025 Jan;104(1):515-525. doi: 10.1007/s00277-024-05958-8. Epub 2024 Sep 4. PMID 39227450
- [Derived] Fu W, Bang SM, Huang H, Kim K, Li W, An G, Lee JJ, Cai Z, Jin J, Wang Y, Lin TL, Chim CS, Qi M, Wang J, Lu X, Song Y, Jia B, Yang X, Liu W, Zhou T, Yin L, Li Y, Zhang R, Hou J, Wang J. Bortezomib, Melphalan, and Prednisone With or Without Daratumumab in Transplant-ineligible Asian Patients With Newly Diagnosed Multiple Myeloma: The Phase 3 OCTANS Study. Clin Lymphoma Myeloma Leuk. 2023 Jun;23(6):446-455.e4. doi: 10.1016/j.clml.2023.02.009. Epub 2023 Mar 4. PMID 37024420